CLINICAL TRIAL: NCT00768391
Title: Phase I Study of Anti-Platelet Derived Growth Factor Receptor Alpha (PDGFRa) Monoclonal Antibody IMC-3G3 in Patients With Advanced Solid Tumors Who No Longer Respond to Standard Therapy or for Whom no Standard Therapy is Available
Brief Title: Study of IMC-3G3 in Patients With Tumors That Are Not Responding to Standard Therapies or No Therapy is Available
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, ImClone LLC
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 13937; CP15-0601 (Other: ImClone, LLC); I5B-IE-JGDC (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-10-06; First posted 2008-10-08 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Solid Tumors
Keywords: Tumors; Lymphoma; Antibodies, Monoclonal
MeSH Terms: conditions — Neoplasms; Lymphoma | interventions — olaratumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMC-3G3 (Experimental): All patients will receive intravenous infusions of IMC-3G3, with the dose depending on which cohort they are enrolled into.
  Interventions: Biological: IMC-3G3

INTERVENTIONS:
Biological: IMC-3G3 — Intravenously, once every week for Cohorts 1 through 3 and once every other week for Cohorts 4 and 5. Starting dose will be 4mg/kg in Cohort 1, with dose doubling between cohorts. Dose escalation of 100% (2 x previous dose) Dose escalation increment reduced to 33% (1.33 x previous dose). Cohorts 4 and 5 will receive 15mg/kg and 20mg/kg, intravenously, once every other week.

SUMMARY:
The purpose of this study is to determine if IMC-3G3 is safe for patients, and also to determine the best dose of IMC-3G3 to give to patients.

DETAILED DESCRIPTION:
The purpose of this study is to establish the safety profile and maximum tolerated dose (MTD) of the anti-PDGFRα monoclonal antibody IMC-3G3 in patients with advanced solid tumors who no longer respond to standard therapy or for whom no standard therapy is available.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathological-documented, measurable, or non measurable, advanced primary tumor or recurrent solid tumor or lymphoma unresponsive to standard therapy or for which there is no standard therapy available.
2. Eastern Cooperative Oncology Group (ECOG) performance status score of ≤ 2 at study entry.
3. Able to provide written informed consent.
4. Age 18 years or older.
5. Life expectancy of > 3 months.
6. Adequate hematologic function, as defined by: an absolute neutrophil count ≥ 1500/mm3; a platelet count ≥ 100,000/mm3
7. Adequate hepatic function, as defined by: a total bilirubin level ≤ 1.5 x the upper limit of normal (ULN); aspartate transaminase (AST) and alanine transaminase (ALT) levels ≤ 2.5 x the ULN or ≤ 5 x the ULN if known liver metastases
8. Adequate renal function, as defined by serum creatinine level ≤ 1.5 x the ULN.
9. Uses effective contraception (per the institutional standard), if procreative potential exists.
10. Adequate recovery from recent surgery, chemotherapy, and radiation therapy.
11. Accessible for treatment and follow-up, must be treated at the participating center.

Exclusion Criteria:

1. Received chemotherapy or therapeutic radiotherapy 28 days prior to the first dose of study medication or has ongoing side effects ≥ grade 2 due to agents administered more than 28 days earlier.
2. Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection requiring parenteral antibiotics; symptomatic congestive heart failure; unstable angina pectoris, angioplasty, stenting, or myocardial infarction 6 months prior to the first dose of study medication; uncontrolled hypertension; clinically significant cardiac arrhythmia including but not limited to: multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia that is symptomatic or requires treatment or asymptomatic sustained ventricular tachycardia; uncontrolled diabetes; psychiatric illness/social situations that would compromise patient safety or limit compliance with study requirements
3. Progressive or symptomatic brain metastases
4. Has a serious or nonhealing active wound, ulcer, or bone fracture.
5. Known human immunodeficiency virus positivity.
6. Major surgical procedure, an open biopsy, or a significant traumatic injury 28 days prior to treatment.
7. Is currently or has recently used (28 days prior to) a thrombolytic agent.
8. Currently using full-dose warfarin (an exception is low-dose warfarin to maintain patency of pre-existing, permanent, indwelling intravenous [I.V.] catheters; for patients receiving warfarin, the international normalized ratio [INR] should be < 1.5). A patient requiring heparin is excluded.
9. Undergoes chronic daily treatment with aspirin (> 325 mg/day) or nonsteroidal anti-inflammatory medications known to inhibit platelet function (cyclooxygenase-2 [COX-2] inhibitors are permitted).
10. Has a history or clinical evidence of a deep venous or arterial thrombosis (including pulmonary embolism) 6 months prior to the first dose of study medication.
11. Has proteinuria ≥ 2+ by routine urinalysis
12. Pregnancy (confirmed by serum beta human chorionic gonadotropin) or lactating
13. Received prior treatment with agents targeting the PDGFR ligand or receptor 6 weeks prior to the first dose of study medication.
14. Received prior treatment with monoclonal antibodies 6 weeks prior to the first dose of study medication.
15. Has a history of allergic reactions to monoclonal antibodies or other therapeutic proteins.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-12; Primary Completion 2009-03 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Summary of Participants Reporting Adverse Events | Approximately 36 months
Maximum Tolerated Dose (MTD) | Approximately 36 months
  After all patients complete a cohort, toxicity data is reviewed before the next cohort of patients is treated at the next higher dose level

SECONDARY OUTCOMES:
Pharmacokinetics | 6 weeks
Anti-IMC-3G3 Antibody Assessment | Approximately 36 months
Antitumor Activity of IMC-3G3 as Monotherapy | 6 weeks
Pharmacodynamics | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: E-mail: ClinicalTrials@ ImClone.com, Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - ImClone Investigational Site, Indianapolis, Indiana
  - ImClone Investigational Site, Houston, Texas